CLINICAL TRIAL: NCT00777608
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial, With Placebo Run-In, and an Open-Label Treatment Period, to Evaluate the Performance of the CogState Computerized Neuropsychological Battery and the ADAS-Cog in Generally Cholinesterase-naive AD Patients
Brief Title: A Study to Test the Performance of the CogState Computerized Neuropsychological Battery in Patients With Alzheimer's Disease (0000-086)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-086; 2008_573
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2011-02-24 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Jogging; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Donepezil 5-10 mg (Experimental): There will be a 14 day period when all participants will receive placebo, followed by 5 mg donepezil, once daily for 14 days then titrated to 10 mg donepezil once daily for 70 days. Participants may then receive open-label donepezil for an additional 24 weeks.
  Interventions: Drug: Comparator: Placebo 5mg (run in); Drug: Donepezil 5 - 10 mg; Drug: Donepezil 10 mg
- Placebo (Placebo Comparator): There will be a 14 day period when all participants will receive placebo. Participants will take placebo capsules orally, once daily for 84 days. Participants may then receive open-label donepezil for an additional 24 weeks.
  Interventions: Drug: Comparator: Placebo 5mg (run in); Drug: Comparator: Placebo 5-10 mg; Drug: Donepezil 10 mg

INTERVENTIONS:
Drug: Comparator: Placebo 5mg (run in) — Matching placebo to donepezil - 5 mg capsules orally for 14 day run in prior to randomization.
Drug: Donepezil 5 - 10 mg — Donepezil 1 capsule (5 mg) orally, once daily for 14 days.
  Donepezil 2 capsules (total 10 mg) once daily for 70 days (days 15-84).
  Arms: Donepezil 5-10 mg
Drug: Comparator: Placebo 5-10 mg — Matching placebo to donepezil, 1 capsule (5 mg) orally, once daily for 14 days.
  Matching placebo to donepezil 2 capsules (total 10 mg) once daily for 70 days (days 15-84).
  Arms: Placebo
Drug: Donepezil 10 mg — Donepezil 2 capsules (total 10 mg) orally, once daily for 24 weeks, from day 85 (optional).

SUMMARY:
This study will evaluate the performance of the CogState computerized neuropsychological battery, Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) and Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) in participants with mild-to-moderate Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Participant is ambulatory, male or female and 55 years of age or older
* Participant has reliable informant/caregiver who can communicate effectively with the study site and personnel

Exclusion Criteria:

* Participant has a history within the last 6 months or current evidence of a psychotic disorder or an active major depressive disorder or participant has any history of schizophrenia
* Participant has a history of multiple and/or serious allergies to drugs or food or a history of an allergic reaction to more than 3 drug classes

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil 5-10 mg: Participants were randomized to donepezil for 84 days
- Placebo: Participants were randomized to placebo for 84 days
Period: Overall Study
Arm/Group | Donepezil 5-10 mg | Placebo
Started | 53 | 53
Completed | 49 | 47
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Investigator Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil 5-10 mg | Placebo | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Customized [Number; unit: Participants] — Age >= 55 years
  Participants | 53 | 53 | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Computer-based Cognitive Assessment (CogState) Composite Score at Week 4
Description: CogState is a simple, brief computerized neuropsychological battery to evaluate cognitive impairments characterizing mild-to-moderate Alzheimer's Disease (AD). The composite CogState assesses attention and memory functions - including Verbal episodic memory, Visual Episodic Memory, Psychomotor function, Visual attention and working memory. CogState scores are measured on a linear scale (with no maximum score) and a reduction in scores compared to baseline indicates an improvement in cognitive functions. Reported here is the change in the CogState Composite Score at Week 4 compared to baseline.
Time Frame: Baseline and 4 weeks
Population: The analysis for the primary and secondary CogState endpoints was done on a per protocol basis (only participants who were compliant and successfully tolerated the forced titration after 2 weeks of treatment were included in the analysis).
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Donepezil 5-10 mg | Placebo
Number analyzed (Participants) | 38 | 43
Score on a scale | -0.10 (0.07) | -0.07 (0.06)
Statistical Analysis 1: Comparison: Donepezil 5-10 mg vs Placebo; Test type: Superiority or Other; p = 0.231, ANOVA; Mean Difference (Final Values) = -0.07, 90% CI 2-sided [-0.2 to 0.08]

2. Secondary Outcome: Evaluate the Efficacy of Donepezil by Determining the Change in Mean CogState Composite Score at Week 2, Week 8 and Week 12
Description: CogState is a simple, brief computerized neuropsychological battery to evaluate cognitive impairments characterizing mild-to-moderate Alzheimer's Disease (AD). The composite CogState assesses attention and memory functions - including Verbal episodic memory, Visual Episodic Memory, Psychomotor function, Visual attention and working memory. CogState scores are measured on a linear scale (no maximum score) and a reduction in scores compared to baseline indicates an improvement in cognitive functions. Reported here is the change from baseline in the CogState Composite Score at Weeks 4, 8 and 12.
Time Frame: Baseline and 2 weeks, 8 weeks and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Donepezil 5-10 mg | Placebo
Number analyzed (Participants) | 38 | 43
Score on a scale
  Week 2 (N=38, N=43) | -0.2 (0.07) | -0.006 (0.06)
  Week 8 (N=38, N=40) | -0.1 (0.07) | -0.02 (0.07)
  Week 12 (N=38, N=41) | -0.2 (0.07) | -0.09 (0.07)
Statistical Analysis 1: Comparison: Donepezil 5-10 mg vs Placebo; Test type: Superiority or Other; p = 0.041, ANOVA; Mean Difference (Final Values) = -0.2, 90% CI 2-sided [-0.3 to -0.008], Standard Error of Mean 0.09 — Statistical analysis for Week 2
Statistical Analysis 2: Comparison: Donepezil 5-10 mg vs Placebo; Test type: Superiority or Other; p = 0.143, ANOVA; Mean Difference (Final Values) = -0.1, 90% CI 2-sided [-0.3 to 0.06], Standard Error of Mean 0.09 — Statistical analysis for Week 8
Statistical Analysis 3: Comparison: Donepezil 5-10 mg vs Placebo; Test type: Superiority or Other; p = 0.226, ANOVA; Mean Difference (Final Values) = -0.07, 90% CI 2-sided [-0.2 to 0.09], Standard Error of Mean 0.10 — Statistical analysis for Week 12

3. Secondary Outcome: Evaluate the Efficacy of Donepezil by Determining the Change in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Score at Week 4, Week 8 and Week 12
Description: The ADAS-Cog is a psychometric instrument that evaluates memory, attention,
  reasoning, language, orientation and praxis using an 11-point AD Assessment Scale. It has a minimum score of 0 and a maximum severity score of 70, and a higher score indicates more impairment. A reduction in scores compared to baseline indicates an improvement in cognitive functions. Reported here is the change in the ADAS-Cog score at Weeks 4, 8 and 12 compared to baseline.
Time Frame: Baseline and 4 weeks, 8 weeks and 12 weeks.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Donepezil 5-10 mg | Placebo
Number analyzed (Participants) | 38 | 43
Score on a scale
  Week 4 (N=38, N=43) | 0.2 (0.8) | -0.3 (0.7)
  Week 8 (N=37, N=40) | 0.07 (1.0) | -0.7 (1.0)
  Week 12 (N=38, N=40) | -1.4 (1.0) | -1.0 (1.0)
Statistical Analysis 1: Comparison: Donepezil 5-10 mg vs Placebo; Test type: Superiority or Other; p = 0.324, ANOVA; Mean Difference (Final Values) = 0.5, 90% CI 2-sided [-1.2 to 2.2], Standard Error of Mean 1.0 — Statistical analysis for Week 4
Statistical Analysis 2: Comparison: Donepezil 5-10 mg vs Placebo; Test type: Superiority or Other; p = 0.285, ANOVA; Mean Difference (Final Values) = 0.8, 90% CI 2-sided [-1.5 to 3.1], Standard Error of Mean 1.4
Statistical Analysis 3: Comparison: Donepezil 5-10 mg vs Placebo; Test type: Superiority or Other; p = 0.401, ANOVA; Mean Difference (Final Values) = -0.3, 90% CI 2-sided [-2.6 to 1.9], Standard Error of Mean 1.3 — Statistical analysis for Week 12

ADVERSE EVENTS:
Groups:
- Donezepil 5-10 mg: Participants were randomized to donepezil for 84 days
Arm/Group | Donezepil 5-10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/53 | 0/53
Other Adverse Events (participants affected / at risk) | 10/53 | 9/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donezepil 5-10 mg (N=53) | Placebo (N=53)
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Donezepil 5-10 mg (N=53) | Placebo (N=53)
Nausea (Gastrointestinal disorders) | 7 | 5
Dizziness (Nervous system disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No